CLINICAL TRIAL: NCT05319561
Title: Dissemination and Implementation of a Videoconference Antimicrobial Stewardship Team (VAST)
Brief Title: Dissemination and Implementation of a Videoconference Antimicrobial Stewardship Team
Acronym: VAST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 20-246; HX003364 (Other Grant/Funding Number: HSR&D)
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Common Infections; Urinary Tract Infections; Pneumonia
Keywords: antimicrobial stewardship; telehealth
MeSH Terms: conditions — Urinary Tract Infections; Pneumonia

STUDY DESIGN:
Intervention Model Description: The Practical, Robust Implementation and Sustainability Model (PRISM) is an expansion of the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) model. Briefly, PRISM expands RE-AIM to further consider key contextual factors related to implementation, evaluation and dissemination of health services programs. The investigators will use PRISM and RE-AIM to inform implementation, evaluation and maintenance of the intervention as the investigators seek to disseminate the VAST beyond the 2 pilot sites
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VAST+ (Experimental): Sites that implement the VAST augmented by quarterly facility-level Antibiotic Use Reports (VAST+).
  Interventions: Other: Antibiotic Use Report
- VAST - (No Intervention): to sites that implement the VAST and do NOT receive a quarterly facility-level Antibiotic Use Reports (VAST-).

INTERVENTIONS:
Other: Antibiotic Use Report — The Antibiotic Use Report uses both text and graphics to communicate successes and improvement opportunities specific to the VAMC for which it is prepared. The graphs summarize overall antibiotic use over the previous year, with additional information regarding use of broad- and narrow-spectrum agents. Further, each Antibiotic Use Report compares or "benchmarks" the individual VAMC for which it is prepared to other VAMCs in the same Medical Complexity Group. This approach adapts and expands peer comparison, which has proven effective at reducing inappropriate antibiotic use in outpatient settings.
  Arms: VAST+

SUMMARY:
Antimicrobial-resistant and healthcare-associated pathogens are a global health threat. The goals of antimicrobial stewardship are to minimize unnecessary and inappropriate antimicrobial use as a means to combat antimicrobial resistance. Previously, the investigators implemented a Videoconference Antimicrobial Stewardship Team (VAST) at 2 VA Medical Centers (VAMCs), using telehealth to connect clinicians at a rural VAMC to a geographically distant infectious disease expert Both VASTs successfully decreased overall antibiotic use in acute and long-term care units. This project will expand the VAST approach to other VAMCs and test the hypothesis that quarterly reports that quantify facility-level antibiotic use will enhance the efficacy of VASTs to support antimicrobial stewardship. This work will directly increase access to antimicrobial stewardship consultation at rural VA facilities, which are often underserved by infectious disease expertise.

DETAILED DESCRIPTION:
Background: Antimicrobial stewardship guidelines call for a multidisciplinary team with an infectious disease (ID) physician and ID-trained clinical pharmacist as core members. Unfortunately, there are insufficient ID-trained specialists to staff on-site antimicrobial stewardship programs throughout VA.

Significance: This proposal is highly significant for Veterans and the goals of VA. Veterans experience many of the risk factors associated with development of antimicrobial resistant and healthcare-associated infections. The unprecedented effects of the novel Coronavirus disease 2019 (COVID-19) on the health of Veterans and on the entire healthcare system makes the demand for ID expertise even more apparent, especially in long-term care. Also, this study directly addresses the VA MISSION ACT to improve access to care, timeliness and quality of care, using telehealth services. Finally, this project is aligned with the priorities of operation partners: VA Antimicrobial Stewardship Taskforce (ASTF), the VA National Infectious Disease Service (NIDS), VA Pharmacy Benefits Management (PBM) Services, and the Office of Rural Health.

Innovation and Impact: The design is innovative because the investigators will systematically test and assess implementation barriers to telehealth for antimicrobial stewardship, a novel approach that has not been implemented in VA facilities, other than in the investigators' previous pilot study. Further, the Antibiotic Use Reports (AURs) are an innovative adaptation of peer-comparison, an antibiotic stewardship strategy successful in outpatient settings. This project will provide findings for a scalable model that could be deployed nationally to all applicable VAMCs, continuing the role of VHA as a leader in implementing large-scale interventions focused on prevention and management of ID and stewardship.

Specific Aims: The goal is to implement a multidisciplinary videoconference antimicrobial stewardship team (VAST) in VAMCs using SCAN-ECHO. The central hypothesis is that feedback reports that quantify facility-level antibiotic use will enhance the efficacy of VASTs to support antimicrobial stewardship. The investigators propose a Type 2 hybrid effectiveness-implementation design, comparing clinical effectiveness in sites that implement the VAST alone (VAST-) to sites that implement the VAST augmented by facility-level Antibiotic Use Reports (VAST+). Aims are: 1) Identify and test effective strategies for implementing the VAST; 2) Determine the influence of the VAST overall and VAST+ on the care of Veterans with suspected infections; 3) Determine the influence of the VAST overall and VAST+ on antibiotic use at each VAMC.

Methodology: The investigators will randomize rural VAMCs that do not have ID-trained professionals on staff to implement the VAST alone (VAST-) versus VAST + antibiotic use feedback (VAST+). Aim 1: The investigators will assess modification and adaptations at the intervention sites and by the infectious disease experts. Methods will include process maps and semi-structured interviews to gather qualitative data about what key VAST members perceive as facilitators, barriers and burden to VAST implementation. The investigators will also evaluate costs of implementation. Aim 2: The investigators will evaluate the Veteran population served, clinical activities, and user perceptions of the VAST. The investigators will assess the concordance of clinical care with recommendations from evidence-based clinical practice guidelines. VAST members' perceptions of the quality and timeliness of care will be evaluated. Aim 3: The primary outcome measure will be overall rates of antibiotic use. Secondary outcomes will be changes in the rates of broad-spectrum antibiotic use, antibiotic starts, and length of antibiotic therapy.

Next steps/Implementation: Testing effective implementation of the VAST at additional VAMCs is an important step toward augmenting antimicrobial stewardship in both acute- and long-term care settings. In collaboration with VA clinical operation partners, outcomes from this trial will be used to roll-out an implementation playbook to be used by other VAMCs, as well as non-VA settings.

ELIGIBILITY:
Inclusion Criteria:

* VA medical centers without local ID expertise that pair with an ID-expert from another VA medical center.

Exclusion Criteria:

* (none)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Days of Antibiotic Therapy / 1000 Bed Days of Care | 2.25 years
  Days of antibiotic therapy per 1000 days of care (DOT/1000 DOC), measures the overall rate of antibiotic use and is a common metric that accounts for dose adjustments, including for people who receive dialysis. Administration of any dose of an antimicrobial on a given day represents a single DOT for that agent, regardless of the number of times the doses are administered or the dose strength.

SECONDARY OUTCOMES:
Rate of broad-spectrum antibiotics | 2.25 years
  The investigators will specifically examine the rate of broad-spectrum antibiotics, defining broad-spectrum agents as those with an Antibiotic Spectrum Index score of 8. This scale ranges from 1 to 13; the ASIs for penicillin, doxycycline, ciprofloxacin, and ertapenem are 2, 5, 8 and 9, respectively.
Antibiotic Starts | 2.25 years
  The investigators will measure the rate of antibiotic starts (new prescriptions), calculated as the number of starts per 1000 DOC. The fourth metric is the length of antibiotic therapy in days. For people on hemodialysis, up to 72 hours may occur between doses of specific agents (e.g. vancomycin, aminoglycosides, several cephalosporins); these will be considered as a single course.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Lynn Paige Jump, MD PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA; Charlesnika Tyon Evans, PhD MPH BS, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (2):
- United States (2):
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Final data sets underlying all publications resulting from the proposed research will not be shared outside VA, except as required under the Freedom of Information Act (FOIA). Reasons for this are (i) the sample size will be too large to obtain informed consents and HIPAA authorizations and (ii) public disclosure of the final study data containing protected health information (PHI) is inconsistent with the IRB approved waiver of informed consent and waiver of HIPAA authorization that will be sought.

REFERENCES:
- [Result] Fabre V, Davis A, Diekema DJ, Granwehr B, Hayden MK, Lowe CF, Pfeiffer CD, Sick-Samuels AC, Sullivan KV, Van Schooneveld TC, Morgan DJ. Principles of diagnostic stewardship: A practical guide from the Society for Healthcare Epidemiology of America Diagnostic Stewardship Task Force. Infect Control Hosp Epidemiol. 2023 Feb;44(2):178-185. doi: 10.1017/ice.2023.5. PMID 36786646

DOCUMENTS (1):
  • Informed Consent Form (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT05319561/ICF_000.pdf